CLINICAL TRIAL: NCT05112484
Title: Importance of Therapeutic Monitoring of Orally Administered Disease-modifying Drugs Used in the Treatment of Multiple Sclerosis
Brief Title: Therapeutic Monitoring of Drugs Used in the Treatment of Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-02/06/2021/2.0; 2021-003195-13 (EudraCT Number)
Record Dates: First submitted 2021-10-13; First posted 2021-11-09 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Therapeutic Drug Monitoring; Concentrations; Disease-Modifying Drugs
MeSH Terms: conditions — Multiple Sclerosis | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The only difference will be the collection of 2 extra tubes for each standard and routine collection from one pre-drug injection and 1 additional tube 2-3 hours after drug administration, either from a new injection or with an established cannula, for a maximum of 3 years (depending on the time of entry into the research project). One blood tube will be taken for genetic testing for the duration of the study, again with standard and routine single injections before taking the drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Gilenya: Gilenya (fingolimod) - first registration 17 March 2011, last renewal 16 November 2020, selective immunosuppressant (ATC code L04AA27), sphingosine-1-phosphate receptor modulator
  Interventions: Diagnostic Test: Measurement of concentrations of orally-used DMDs; Diagnostic Test: Genetic testing; Diagnostic Test: Parameters for routine use of DMDs; Other: Side effects of orally used DMDs
- Tecfidera: Tecfidera (dimethyl fumarate) - first registration 30 January 2014, last renewal 20 September 2018, cytostatic and immunomodulatory drug (ATC code L04AX07), an activator of the transcription pathway of nuclear factor Nrf2
  Interventions: Diagnostic Test: Measurement of concentrations of orally-used DMDs; Diagnostic Test: Genetic testing; Diagnostic Test: Parameters for routine use of DMDs; Other: Side effects of orally used DMDs
- Mavenclad: Mavenclad (cladribine) - first registration 22/08/2017, selective immunosuppressant (ATC code L04AA40), nucleoside analogue of deoxyadenosine
  Interventions: Diagnostic Test: Measurement of concentrations of orally-used DMDs; Diagnostic Test: Genetic testing; Diagnostic Test: Parameters for routine use of DMDs; Other: Side effects of orally used DMDs
- Aubagio: Aubagio (teriflunomide) - first registration on 26 August 2013, last renewal on 28 May 2018, selective immunosuppressant (ATC code L04AA31), an inhibitor of the mitochondrial enzyme dihydroorotate dehydrogenase
  Interventions: Diagnostic Test: Measurement of concentrations of orally-used DMDs; Diagnostic Test: Genetic testing; Diagnostic Test: Parameters for routine use of DMDs; Other: Side effects of orally used DMDs

INTERVENTIONS:
Diagnostic Test: Measurement of concentrations of orally-used DMDs — For effectiveness - the measured concentrations of orally used "DMDs" will be correlated with the clinical condition of patients with MS (usual clinical examinations such as physical assessment of clinical condition, evaluation of EDSS scale, MSQOL-54 quality of life questionnaire, and routine magnetic resonance imaging of the brain once a year). At the same time, the relationship between the measured concentrations of orally used "DMDs" and the concentrations of other biomarkers of MS, such as signs of axonal (so-called plasma neurofilament light chain - "pNfL") and glial (so-called chitinase 3-like 1 - "CHI3L1") damage, will be analyzed. concentrations of selected cytokines, concentrations of CD4 + and CD8 + T-lymphocytes, and the results of a genetic examination of drug transporters, again with an effect on the clinical condition of the patient.
Diagnostic Test: Genetic testing — One blood tube will be taken for genetic testing for the duration of the study, again with standard and routine single injections before taking the drug.
Diagnostic Test: Parameters for routine use of DMDs — For safety - the usual parameters for routine use of "DMDs" will be monitored (blood count, liver tests, renal function, etc. according to the specifics of individual drugs).
Other: Side effects of orally used DMDs — For tolerability - possible side effects of orally used "DMDs" will be monitored and the effect of genetic testing of drug transporters will be analyzed.

SUMMARY:
The main goal of multiple sclerosis (MS) treatment is to prevent further relapses of the disease and the progression of neurological deficit. Although MS cannot yet be cured, early control of symptoms and reduction of disease progression is associated with a longer time to disability and improve long-term treatment outcomes. Currently, MS is treated using a multidisciplinary approach, which consists of treatment with so-called "disease-modifying drugs" ("DMDs"), symptomatic therapy of individual symptoms, lifestyle adjustments, psychological support, and rehabilitation interventions. According to the latest results, treatment with "DMDs" can reduce the annual incidence of relapses by 29-68% compared to placebo or an active comparator. Thus, as can be seen, even this group of modern drugs does not completely compensate for MS in many patients. For this reason, there is a need to use certain parameters to best assess the effectiveness of individual treatments in specific patients with MS in routine clinical practice. Therapeutic drug monitoring (TDM) is a specific method of clinical pharmacology that has long been used to monitor therapy for a variety of diseases by measuring drug concentrations in body fluids (plasma, serum, whole blood, cerebrospinal fluid, breast milk) with subsequent interpretation by clinical pharmacologist and acceptance by the clinician. The groups of drugs for which TDM is routinely performed include selected groups of antibiotics (aminoglycosides, vancomycin, beta-lactams), immunosuppressants, digoxin, and especially drugs used in neurology and psychiatry (antiepileptics and psychotropic drugs). As far as "DMDs" is concerned, the first data on the possibility of using TDM in the therapy of MS have already appeared in the professional literature, but these are so far rare and completely insufficient. In addition, individual drugs differ not only in efficacy but also in dose, dosing schedule, and safety profile. The development of new analytical methods to determine serum or whole blood "DMDs" concentrations, together with the objectification of the relationship between measured concentrations to the patient's clinical condition and the possibility of objectifying patient adherence to treatment, could therefore significantly help individualize the dosage of "DMDs" in each individual patient.

DETAILED DESCRIPTION:
The study group will consist of individuals with MS who will be indicated for some of the orally used disease-modifying drugs ("DMDs") - fingolimod, dimethyl fumarate, cladribine, or teriflunomide, both patients with established treatment and patients who will have this medication newly used. All medical care will be performed according to the habits and decisions of the attending physician depending on the clinical condition of the patient, in addition, only 3 blood tubes will be taken on the day of scheduled standard collection and 1 blood tube for the entire duration of the study for genetic testing. Of these, 2 tubes will be collected as part of a standard fasting sample from fasting before drug administration with other routinely collected blood samples (including one tube for the duration of the genetic testing study) and 1 tube will be collected 2-3 hours after drug administration. to determine the maximum drug concentration. For the patient, all the load will mean only one extra collection, ie a collection after taking the drug, either from a new injection or with an inserted cannula. Blood samples obtained from 2 tubes taken on an empty stomach will be used to determine the concentration of "DMDs" of the drug before use and to analyze other biomarkers that could be used to evaluate the patient's clinical condition, such as signs of axonal damage (plasma neuro-filament light chain - pNfL). "), Glial damage (so-called chitinase 3-like 1 -" CHI3L1 "), concentrations of selected cytokines or concentrations of CD4 + and CD8 + T cells. One tube of blood taken also on an empty stomach, once for the duration of the study, will be used for genetic testing of drug transporters such as P-gp (ABCB1) or BCRP (ABCG2). At the same time, the patient will perform the usual clinical examinations (physical assessment of the clinical condition, evaluation of the EDSS scale, monitoring of possible side effects of the medication used and the MSQOL-54 quality of life questionnaire) and once a year routine magnetic resonance imaging of the brain. The information thus obtained will be correlated with the achieved concentration of "DMDs" used to determine whether this group of drugs would be suitable for routine therapeutic monitoring, similar to antiepileptics, for which TDM has been part of routine clinical practice to optimize since the 1970s. pharmacotherapy in individual patients to compensate for the clinical condition with minimal side effects. The investigators would also try to establish a reference range of individual "DMDs", which would be defined as the concentration of drug in serum or whole blood at which most patients are expected to achieve an optimal clinical response. However, since some patients may (similarly to antiepileptics) require a concentration outside this reference range, the investigators would try to determine the so-called "individual therapeutic concentration" in these cases, i.e. the concentration at which MS without an MS attack with good tolerability of medication would be achieved, possibly as the best compromise between improving MS control and concentration-dependent side effects. For the patient, all loading will mean only one extra collection, i.e. a post-drug collection, which can be done either from a new injection or with an inserted cannula. This collection may involve common risks, such as bleeding from an injection site due to insufficient compression of the injection site, the development of a hematoma, or a drop in blood pressure. By obtaining the valuable parameters mentioned above, not only others, resp. future patients with MS, but due to the short duration of the study and at the same time the lifelong influence of the patient with multiple sclerosis, these results may help to optimize the pharmacotherapy of "DMDs" also in a specific individual patient - study participant. However, because long-term patient adherence to treatment is equally important for MS compensation, the introduction of TDM "DMDs" for attending physicians could help not only to optimize the pharmacotherapy of MS but also to control the patient's adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with MS of all forms using any of the oral "DMDs"
* men and women older than 18 years
* signature of the Informed Consent to Participate in the Study

Exclusion Criteria:

* minor patients (below 18 years of age)
* refusal to sign the Informed Consent to Participate in the Study
* refusal of blood samples taken beyond standard examinations

Criteria for exclusion from the study

* non-compliance with the treatment regimen according to the decision of the attending physician
* non-participation in blood samples taken as part of standard examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants of all four study groups will be both patients with established treatment and patients who will be newly introduced to the "DMDs" medication.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Correlation of measured concentrations of orally used "DMDs" with the clinical condition of patients with MS | up to 3 years
  Correlation of measured concentrations of orally used "DMDs" with the clinical condition of patients with MS will be observed.
Objectification of adherence to treatment in individual "DMDs" | up to 3 years
  Objectification of adherence to treatment in individual "DMDs" will be observed.
The percentage of patients with "DMDs" in whom therapeutic monitoring is used | up to 3 years
  The percentage of patients with "DMDs" in whom therapeutic monitoring is used will be observed.

SECONDARY OUTCOMES:
Analysis of the relationship between the measured concentrations of orally used "DMDs" and the concentrations of other biomarkers of MS | up to 3 years
  Analysis of the relationship between the measured concentrations of orally used "DMDs" and the concentrations of other biomarkers of MS, such as signs of axonal (so-called plasma neurofilament light chain - "pNfL") and glial (so-called chitinase 3-like 1 - "CHI3L1") damage, concentrations of selected cytokines, concentrations of CD4 + and CD8 + T-lymphocytes
Analysis of the relationship between the measured concentrations of orally used "DMDs" with the results of genetic examination of drug transporters of the P-gp (ABCB1) and BCRP (ABCG2) type | up to 3 years
  analysis of the relationship between the measured concentrations of orally used "DMDs" with the results of genetic examination of drug transporters of the P-gp (ABCB1) and BCRP (ABCG2) type

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Kacířová, Assoc. Prof.,MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - University of Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Hunter SF. Overview and diagnosis of multiple sclerosis. Am J Manag Care. 2016 Jun;22(6 Suppl):s141-50. PMID 27356023
- [Background] McGinley MP, Goldschmidt CH, Rae-Grant AD. Diagnosis and Treatment of Multiple Sclerosis: A Review. JAMA. 2021 Feb 23;325(8):765-779. doi: 10.1001/jama.2020.26858. PMID 33620411
- [Background] Hocevar K, Ristic S, Peterlin B. Pharmacogenomics of Multiple Sclerosis: A Systematic Review. Front Neurol. 2019 Feb 26;10:134. doi: 10.3389/fneur.2019.00134. eCollection 2019. PMID 30863357
- [Background] Grossman I, Knappertz V, Laifenfeld D, Ross C, Zeskind B, Kolitz S, Ladkani D, Hayardeny L, Loupe P, Laufer R, Hayden M. Pharmacogenomics strategies to optimize treatments for multiple sclerosis: Insights from clinical research. Prog Neurobiol. 2017 May;152:114-130. doi: 10.1016/j.pneurobio.2016.02.001. Epub 2016 Mar 4. PMID 26952809
- [Background] Nicholas JA, Edwards NC, Edwards RA, Dellarole A, Grosso M, Phillips AL. Real-world adherence to, and persistence with, once- and twice-daily oral disease-modifying drugs in patients with multiple sclerosis: a systematic review and meta-analysis. BMC Neurol. 2020 Jul 14;20(1):281. doi: 10.1186/s12883-020-01830-0. PMID 32664928
- [Background] Apostolopoulos V, Matsoukas J. Advances in Multiple Sclerosis Research-Series I. Brain Sci. 2020 Oct 29;10(11):795. doi: 10.3390/brainsci10110795. PMID 33137992
- [Background] Jalkh G, Abi Nahed R, Macaron G, Rensel M. Safety of Newer Disease Modifying Therapies in Multiple Sclerosis. Vaccines (Basel). 2020 Dec 26;9(1):12. doi: 10.3390/vaccines9010012. PMID 33375365
- [Background] Madden MC, Vender RL, Friedman M. Effect of hypoxia on prostacyclin production in cultured pulmonary artery endothelium. Prostaglandins. 1986 Jun;31(6):1049-62. doi: 10.1016/0090-6980(86)90208-x. PMID 3094092
- [Background] Rotstein D, Montalban X. Reaching an evidence-based prognosis for personalized treatment of multiple sclerosis. Nat Rev Neurol. 2019 May;15(5):287-300. doi: 10.1038/s41582-019-0170-8. PMID 30940920
- [Background] Olsson A, Gustavsen S, Hasselbalch IC, Langkilde AR, Sellebjerg F, Oturai AB, Sondergaard HB. Biomarkers of inflammation and epithelial barrier function in multiple sclerosis. Mult Scler Relat Disord. 2020 Nov;46:102520. doi: 10.1016/j.msard.2020.102520. Epub 2020 Sep 19. PMID 32980645
- [Background] Hiemke C, Bergemann N, Clement HW, Conca A, Deckert J, Domschke K, Eckermann G, Egberts K, Gerlach M, Greiner C, Grunder G, Haen E, Havemann-Reinecke U, Hefner G, Helmer R, Janssen G, Jaquenoud E, Laux G, Messer T, Mossner R, Muller MJ, Paulzen M, Pfuhlmann B, Riederer P, Saria A, Schoppek B, Schoretsanitis G, Schwarz M, Gracia MS, Stegmann B, Steimer W, Stingl JC, Uhr M, Ulrich S, Unterecker S, Waschgler R, Zernig G, Zurek G, Baumann P. Consensus Guidelines for Therapeutic Drug Monitoring in Neuropsychopharmacology: Update 2017. Pharmacopsychiatry. 2018 Jan;51(1-02):e1. doi: 10.1055/s-0037-1600991. Epub 2018 Feb 1. No abstract available. PMID 29390205
- [Background] Hopkins AM, O'Doherty CE, Foster DJ, Upton RN, Proudman SM, Wiese MD. Individualization of leflunomide dosing in rheumatoid arthritis patients. Per Med. 2014 Jun;11(4):449-461. doi: 10.2217/pme.14.23. PMID 29783485
- [Background] Zarzuelo Romero MJ, Perez Ramirez C, Carrasco Campos MI, Sanchez Martin A, Calleja Hernandez MA, Ramirez Tortosa MC, Jimenez Morales A. Therapeutic Value of Single Nucleotide Polymorphisms on the Efficacy of New Therapies in Patients with Multiple Sclerosis. J Pers Med. 2021 Apr 23;11(5):335. doi: 10.3390/jpm11050335. PMID 33922540
- [Background] Yao X, Wu Y, Jiang J, Chen X, Liu D, Hu P. A population pharmacokinetic study to accelerate early phase clinical development for a novel drug, teriflunomide sodium, to treat systemic lupus erythematosus. Eur J Pharm Sci. 2019 Aug 1;136:104942. doi: 10.1016/j.ejps.2019.05.020. Epub 2019 May 30. PMID 31154006
- [Background] Fewings NL, Gatt PN, McKay FC, Parnell GP, Schibeci SD, Edwards J, Basuki MA, Goldinger A, Fabis-Pedrini MJ, Kermode AG, Manrique CP, McCauley JL, Nickles D, Baranzini SE, Burke T, Vucic S, Stewart GJ, Booth DR. The autoimmune risk gene ZMIZ1 is a vitamin D responsive marker of a molecular phenotype of multiple sclerosis. J Autoimmun. 2017 Mar;78:57-69. doi: 10.1016/j.jaut.2016.12.006. Epub 2017 Jan 4. PMID 28063629
- [Background] Carlstrom KE, Ewing E, Granqvist M, Gyllenberg A, Aeinehband S, Enoksson SL, Checa A, Badam TVS, Huang J, Gomez-Cabrero D, Gustafsson M, Al Nimer F, Wheelock CE, Kockum I, Olsson T, Jagodic M, Piehl F. Therapeutic efficacy of dimethyl fumarate in relapsing-remitting multiple sclerosis associates with ROS pathway in monocytes. Nat Commun. 2019 Jul 12;10(1):3081. doi: 10.1038/s41467-019-11139-3. PMID 31300673
- [Background] Hermann R, Karlsson MO, Novakovic AM, Terranova N, Fluck M, Munafo A. The Clinical Pharmacology of Cladribine Tablets for the Treatment of Relapsing Multiple Sclerosis. Clin Pharmacokinet. 2019 Mar;58(3):283-297. doi: 10.1007/s40262-018-0695-9. PMID 29987837
- [Background] Abdelhak A, Huss A, Stahmann A, Senel M, Krumbholz M, Kowarik MC, Havla J, Kumpfel T, Kleiter I, Wustinger I, Zettl UK, Schwartz M, Roesler R, Friede T, Ludolph AC, Ziemann U, Tumani H. Explorative study of emerging blood biomarkers in progressive multiple sclerosis (EmBioProMS): Design of a prospective observational multicentre pilot study. Contemp Clin Trials Commun. 2020 May 19;18:100574. doi: 10.1016/j.conctc.2020.100574. eCollection 2020 Jun. PMID 32478196
- See also: The Atlas of Multiple Sclerosis — http://www.atlasofms.org